CLINICAL TRIAL: NCT03946358
Title: A Phase II Study Evaluating the Interest to Combine UCPVax a CD4 TH1-inducer Cancer Vaccine and Atezolizumab for the Treatment of Human PapillomaVirus Positive Cancers
Brief Title: Combination of UCPVax Vaccine and Atezolizumab for the Treatment of Human Papillomavirus Positive Cancers (VolATIL)
Acronym: VolATIL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Roche Pharma AG (Industry); National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P/2019/418
Record Dates: First submitted 2019-05-07; First posted 2019-05-10 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck; Anal Canal Cancer; Cervical Cancer
Keywords: Human PapillomaVirus (HPV); Atezolizumab; Cancer vaccine; Cancer immunotherapy; Telomerase
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Anal Canal Carcinoma; Uterine Cervical Neoplasms | interventions — atezolizumab; Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Atezolizumab and UCPVax (Experimental): Induction phase:
  * Atezolizumab 1200 mg intravenous (IV) every 3 weeks since day 1
  * UCPVax (combined with Montanide ISA51 as adjuvant) at 1 mg subcutaneously in two separate sites (one site per peptide) at day 1, 8, 15, 29, 36 and 43 (induction phase).
  Boost phase:
  * UCPVax boosts vaccine every 6 weeks for the 2 first boosts (boost 1 and boost 2) and then every 9 weeks (boost 3 to boost 5)
  * Atezolizumab 1200 mg IV every 3 weeks until disease progression or unacceptable toxicity until disease progression or unacceptable toxicity.
  Interventions: Biological: Blood sample collection; Procedure: Tumor biopsies; Other: CT scan; Drug: Atezolizumab; Drug: UCPVax

INTERVENTIONS:
Biological: Blood sample collection — Four blood samples will be collected at:
  * baseline
  * 2 months from inclusion (+/- 1 week)
  * 4 months from inclusion (+/- 1 week)
  * the end of vaccination visit (+/- 1 week).
  A total of 8 EDTA (ethylenediaminetetraacetic acid) tubes of 6 ml will be collected at each time point to perform:
  PBMC collection: 6 EDTA tubes of 6 ml of peripheral blood mononuclear cell [PBMC] will be sent to the central laboratory (Biomonitoring Platform of Besançon, CHRU de Besançon located at Etablissement Français du Sang) at room temperature within 24 hours via an approved carrier for their processing, storage and immunomonitoring analysis. A sending sheet of the samples will be attached to each single sample.
  Plasma collection: One 6 ml EDTA tube should be frozen in each investigation center for plasma collection.
  Plasma for circulating tumoral DNA (ctDNA) collection: One 6 ml EDTA tube should be frozen in each investigation center for ctDNA collection.
Procedure: Tumor biopsies — A tumor biopsy will be realized and centralized at baseline and at 2 months. Collection of tumor biopsies will be guided by ultrasound or CT scan
Other: CT scan — A CT scan will be planned
  * at baseline
  * at tumor evaluation visit (8 weeks)
  * every 8 weeks (+/- 1 week)
  * at end of treatment visit.
Drug: Atezolizumab — Induction phase: Atezolizumab 1200 mg intravenous every 3 weeks since day 1
  Boost phase: Atezolizumab 1200 mg intravenous every 3 weeks until disease progression or unacceptable toxicity until disease progression or unacceptable toxicity.
  Other Names: anti-PD-L1
Drug: UCPVax — Induction phase: UCPVax (combined with Montanide ISA51 as adjuvant) at 1 mg subcutaneously in two separate sites (one site per peptide) at day 1, 8, 15, 29, 36 and 43 (induction phase).
  Boost phase: UCPVax boosts vaccine every 6 weeks for the 2 first boosts (boost 1 and boost 2) and then every 9 weeks (boost 3 to boost 5).
  Other Names: Vaccine

SUMMARY:
70% all cases of cervical cancer, 95% of anal cancers and about 70% of oropharyngeal cancers are linked to Human Papillomavirus (HPV) infection. HPV oncogenic proteins are trans-activators of telomerase. Indeed, E6 oncoprotein transactivates the human telomerase (hTert). Our group has conducted a clinical trial (NCT02402842) in advanced squamous cell anal cancer (SCCA) and investigators have shown a correlation between the presence of anti-HPV immunity and anti-telomerase T helpher 1 (TH1) CD4 T cell responses, establishing telomerase as an appropriate antigen in HPV-related cancers.

Tumor-reactive CD4+ T cells have been found to ensure efficient effector Cytotoxic T Lymphocytes (CTL) recruitment at the tumor site. Promoting tumor specific TH1 CD4 activation might be an attractive therapeutic option to enhance anti-PD-1/PD-L1 (Programmed cell Death-1/Programmed cell Death-Ligand1) efficacy. However, no option is currently available to expand tumor specific TH1 lymphocytes in most patients. Then, investigators have identified four novel MHC (Major Histocompatibility Complex) class II-restricted peptides derived from human telomerase reverse transcriptase (TERT) referred as "Universal Cancer Peptides" (UCP). UCPVax is a therapeutic cancer vaccine developed by our team and composed of two separate peptides called UCP2 and UCP4 derived from telomerase. This UCPVax vaccine is currently evaluated in a multicenter phase I/II study in Non Small Lung Cancer (NSCLC) (NCT2818426) and seems to show to be safe and immunogenic.

PD-1/PD-L1 immune checkpoint is a relevant candidate target for immunotherapy in HPV+ cancers, based on the prominent role of PD-1 and its ligand PD-L1 in HPV-driven immune-evasion. There is a strong rational of using PD-1 therapy in HPV+ cancers, however anti-PD-1/PD-L1 treatment induces a limited number of long term responses in HPV disease. Combining anti-PD-1/PD-L1 therapy with an antitumor vaccine gains serious consideration in HPV+ cancers. Indeed, anti-cancer vaccines can induce tumor-specific T cells expansion and activation and therefore restore the cancer-immunity cycle in patients lacking pre-existing anti-tumor responses.

So investigators propose to determine the clinical interest and immunological efficacy of a treatment combining the CD4 helper T-inducer cancer vaccine (UCPVax) with atezolizumab in patients with HPV+ cancers by evaluation of the objective response rate at 4 months according to iRecist criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent
2. Histologically confirmed HPV+ cancers, defined by p16+ (IHC) or HPV genotyping, corresponding to one of the following selected squamous cell carcinoma types:

   * Anal cancer
   * Head and Neck carcinoma,
   * cervical and vulvar carcinoma
3. Locally advanced or metastatic disease
4. Pre-treated with at least 1 line of anticancer standard treatment (chemotherapy, radiochemotherapy or targeted therapy…)
5. Age ≥ 18 and ≤ 75 years old
6. Measurable disease defined according to iRECIST v1.1 guidelines (Note: Previously irradiated lesions can be considered as measurable disease only if disease progression has been unequivocally documented at that site since radiation.)
7. Patients must have a mandatory treatment-free interval of at least 21 days following previous systemic anti-cancer treatments
8. Patients who have received previous systemic anticancer treatment and/or radiotherapy should have recovered from any treatment related toxicity, to a level of ≤ grade 1 (according to National Cancer Institute [NCI] common terminology criteria for adverse events, version 5 (CTCAE v5) with the exception of Grade 2 alopecia
9. Performance status < 2 (Annex 3)
10. Availability of a pre-treatment tumor sample (archival FFPE [formalin-fixed paraffin-embedded] block) and presence of a tumor lesion suitable for a biopsy
11. Patient affiliated to or beneficiary of French social security system
12. Ability to comply with the study protocol, in the Investigator's judgment.

Exclusion Criteria:

Non-eligible to a clinical trial:

1. Patients previously exposed to anti-tumor immunotherapy as anti-PD-1, anti-PD-L1, or anti-CTLA4 agent or any immune therapy. (HPV vaccination is allowed)
2. Diagnosis of additional malignancy within 3 years prior to the inclusion with the exception of curatively treated basal cell carcinoma of the skin and/or curatively resected in situ cervical or breast cancer
3. Patient with any medical or psychiatric condition or disease, which would make the patient inappropriate for entry into this study
4. Current participation in a study of an investigational agent or in the period of exclusion
5. Pregnancy, breast-feeding or absence/refusal of adequate contraception for fertile patients during the period of treatment and for 6 months from the last treatment administration
6. Patient under guardianship, curatorship or under the protection of justice

   Cancer-specific exclusion criteria:
7. Uncontrolled pleural effusion, pericardial effusion, ascites or symptomatic fistula
8. Uncontrolled tumor-related pain: exposing patients to risk of exposure to corticoids or iterative hospitalizations. Symptomatic lesions amenable to palliative radiotherapy should be treated prior to randomization. Patients should be recovered from the effects of radiation. There is no required minimum recovery period
9. Known active central nervous system metastases and/or carcinomatous meningitis. Subject with previously treated brain metastases and with radiological and clinical stability are allowed

   Non-eligible to treatment:
10. Inadequate organ functions: known cardiac failure of unstable coronaropathy, respiratory failure, or uncontrolled infection or another life-risk condition
11. Active or chronic hepatitis B or C and/or HIV positive (HIV 1/2 antibodies patients), or a known history of active Tuberculosis bacillus
12. Any immunosuppressive therapy (i.e. corticosteroids >10mg of hydrocortisone or equivalent dose) within 14 days before the planned start of study therapy
13. Active autoimmune disease that has required a systemic treatment in past 2 years (i.e. corticosteroids or immunosuppressive drugs). Replacement therapy (e.g. thyroxine, insulin) is allowed

    Active or history of autoimmune disease or immune deficiency, including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis, (see Annex 5 for a more comprehensive list of autoimmune diseases and immune deficiencies) with the following exceptions:
    * Patients with a history of autoimmune-related hypothyroidism who are on thyroid replacement hormone are eligible for the study,
    * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study,
    * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:

      1. Rash must cover < 10% of body surface area,
      2. Disease is well controlled at baseline and requires only low-potency topical corticosteroids,
      3. No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high potency or oral corticosteroids within the previous 12 months,
14. Prior allogeneic bone marrow transplantation or prior solid organ transplantation
15. History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
16. Known hypersensitivity or allergy to Chinese hamster ovary cell products or any component of atezolizumab formulation
17. History of idiopathic or secondary pulmonary fibrosis (History of radiation pneumonitis in the radiation field fibrosis is permitted), or evidence of active pneumonitis requiring a systemic treatment with 28 days before the planned start of study therapy
18. Major surgical procedure other than for diagnosis within 4 weeks prior to initiation of study treatment, or anticipation of need for a major surgical procedure during the course of the study
19. Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia
20. Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment. Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study
21. Patients under chronic treatment with systemic corticoids or other immunosuppressive drugs (prednisone or prednisolone ≤ 10 mg/day is allowed) for a period of at least 4 weeks and whose treatment was not stopped 1 week prior to the start of the study treatment
22. Patient with intra-alveolar hemorrhage, pulmonary fibrosis, or uncontrolled asthma, or chronic obstructive disease (COPD), defined as at least 1 hospitalization within 4 months prior to enrollment or as at least 3 exacerbations during the last year prior to enrollment
23. Patients requiring oxygen therapy
24. Patients with LEVF (Left Ejection Ventricular Fraction) <40%
25. Hospitalization for cardiovascular or pulmonary disease within 4 weeks prior to enrollment.
26. Receipt of a live, attenuated vaccine within 4 weeks prior to randomization or anticipation that such a live, attenuated vaccine will be required during the study Note: Patients must agree not to receive live, attenuated influenza vaccine (e.g.,FluMist®) within 28 days prior to randomisation, during treatment or within 5 months following the last dose of atezolizumab
27. Inadequate hematology function: Lymphocyte count at baseline < 800/mm3 ; neutrophil count <1500/mm3, platelets <100000/mm3, Hemoglobin<9g/dL
28. Inadequate hepatic function: bilirubin 2.5 fold ULN (upper limit of normal), AST/ALT (ASpartate Transaminase /ALanine Transaminase) 2.5 fold ULN or 5 fold ULN with liver metastasis, International normalized thromboplastin time ratio >1.5
29. Inadequate renal function: MDRD (Modification of Diet in Renal Disease ) CrCl (Creatinine Clearance) <40ml/min
30. Others inadequate laboratory values: serum albumin<30 g/L; troponin > ULN ; BNP (Brain-Type Natriuretic Peptide) > ULN.
31. Active alcohol or drug abuse.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-02-18 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Objective response rate at 4 months | 4 months
  The main objective of this clinical trial is to assess the efficacy of a strategy combining UCPVax and atezolizumab treatment in patients with HPV+ cancer by evaluation of the objective response rate at 4 months according to iRecist.

SECONDARY OUTCOMES:
Overall survival | through study completion, an average of 2 years
  Delay from the date of inclusion to death from any cause
Progression free-survival | through study completion, an average of 2 years
  Delay from the date of inclusion to the disease progression or death from any cause whichever occurs first
Health related quality of life (HrQoL) | From to inclusion patient for maximum of 2 years
  Health related quality of life will be assessed using EORTC (European Organisation for Research and Treatment of Cancer) questionnaire
Safety of UCPVax in association with anti-PD-L1 | From to inclusion patient for maximum of 2 years
  Toxicities graded according to NCI-CTCAE criteria version 5

CONTACTS AND LOCATIONS:
Overall Officials: Christophe BORG, Pr, Principal Investigator — CHU Besançon
Locations (4):
- France (4):
  - CHU de Besançon, Besançon
  - Centre Georges François Leclerc, Dijon
  - Centre Léon Bérard, Lyon
  - Hospices Civils de Lyon, Lyon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim S, Francois E, Andre T, Samalin E, Jary M, El Hajbi F, Baba-Hamed N, Pernot S, Kaminsky MC, Bouche O, Desrame J, Zoubir M, Ghiringhelli F, Parzy A, De La Fouchardiere C, Smith D, Deberne M, Spehner L, Badet N, Adotevi O, Anota A, Meurisse A, Vernerey D, Taieb J, Vendrely V, Buecher B, Borg C. Docetaxel, cisplatin, and fluorouracil chemotherapy for metastatic or unresectable locally recurrent anal squamous cell carcinoma (Epitopes-HPV02): a multicentre, single-arm, phase 2 study. Lancet Oncol. 2018 Aug;19(8):1094-1106. doi: 10.1016/S1470-2045(18)30321-8. Epub 2018 Jul 2. PMID 30042063
- [Background] Godet Y, Fabre E, Dosset M, Lamuraglia M, Levionnois E, Ravel P, Benhamouda N, Cazes A, Le Pimpec-Barthes F, Gaugler B, Langlade-Demoyen P, Pivot X, Saas P, Maillere B, Tartour E, Borg C, Adotevi O. Analysis of spontaneous tumor-specific CD4 T-cell immunity in lung cancer using promiscuous HLA-DR telomerase-derived epitopes: potential synergistic effect with chemotherapy response. Clin Cancer Res. 2012 May 15;18(10):2943-53. doi: 10.1158/1078-0432.CCR-11-3185. Epub 2012 Mar 8. PMID 22407833
- [Background] Dosset M, Godet Y, Vauchy C, Beziaud L, Lone YC, Sedlik C, Liard C, Levionnois E, Clerc B, Sandoval F, Daguindau E, Wain-Hobson S, Tartour E, Langlade-Demoyen P, Borg C, Adotevi O. Universal cancer peptide-based therapeutic vaccine breaks tolerance against telomerase and eradicates established tumor. Clin Cancer Res. 2012 Nov 15;18(22):6284-95. doi: 10.1158/1078-0432.CCR-12-0896. Epub 2012 Oct 2. PMID 23032748
- [Background] Dosset M, Vauchy C, Beziaud L, Adotevi O, Godet Y. Universal tumor-reactive helper peptides from telomerase as new tools for anticancer vaccination. Oncoimmunology. 2013 Mar 1;2(3):e23430. doi: 10.4161/onci.23430. PMID 23802085
- [Derived] Rebucci-Peixoto M, Vienot A, Adotevi O, Jacquin M, Ghiringhelli F, de la Fouchardiere C, You B, Maurina T, Kalbacher E, Bazan F, Meynard G, Clairet AL, Fagnoni-Legat C, Spehner L, Bouard A, Vernerey D, Meurisse A, Kim S, Borg C, Mansi L. A Phase II Study Evaluating the Interest to Combine UCPVax, a Telomerase CD4 TH1-Inducer Cancer Vaccine, and Atezolizumab for the Treatment of HPV Positive Cancers: VolATIL Study. Front Oncol. 2022 Jul 19;12:957580. doi: 10.3389/fonc.2022.957580. eCollection 2022. PMID 35928870